CLINICAL TRIAL: NCT05818553
Title: A Phase 2,Double-Blind,Randomized Clinical Trial to Explore the Safety,Tolerability,Efficacy, and Pharmacokinetics of PRAX-562 in Pediatric Participants With Developmental and Epileptic Encephalopathies Followed by Open-Label Extension(OLE)
Brief Title: A Clinical Trial of PRAX-562 in Subjects With Developmental and Epileptic Encephalopathies (DEE)
Acronym: EMBOLD
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRAX-562-221
Record Dates: First submitted 2023-03-17; First posted 2023-04-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-01

CONDITIONS: SCN2A Encephalopathy; SCN8A Encephalopathy
Keywords: Pediatric epilepsy; NaV1.2 Voltage-Gated Sodium Channel; SCN2A variant; SCN8A variant; Developmental and epileptic encephalopathy

STUDY DESIGN:
Intervention Model Description: Parallel group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Randomized, Double-Blind 0.5mg/kg/day PRAX-562 or PRAX-562/Placebo (Experimental): Eligible participants from each cohort will be randomized in a 1:1 ratio to either 0.5 milligrams/kilograms/day (mg/kg/day) PRAX-562 for 16 weeks (PRAX-562 arm) or 0.5 mg/kg/day PRAX-562 for 12 weeks and matching placebo for 4 weeks (PRAX-562/placebo arm) administered orally or via gastrostomy tube (G-tube).
  Interventions: Drug: PRAX-562
- Part B: Open-Label Extension Treatment 0.5mg/kg/day PRAX-562 (Experimental): Eligible participants will receive 0.5mg/kg/day administered orally or via G-tube for up to 144 weeks.
  Interventions: Drug: PRAX-562
- Part A: Randomized, Double-Blind 1.0 mg/kg/day PRAX-562 or PRAX-562/Placebo (Experimental): Eligible participants from each cohort will be randomized in a 1:1 ratio to either 1.0 milligrams/kilograms/day (mg/kg/day) PRAX-562 for 16 weeks (PRAX-562 arm) or 1.0 mg/kg/day PRAX-562 for 12 weeks and matching placebo for 4 weeks (PRAX-562/placebo arm) administered orally or via gastrostomy tube (G-tube).
  Interventions: Drug: PRAX-562
- Open-Label Extension Treatment 1.0 mg/kg/day PRAX-562 (Experimental): Eligible participants will receive 1.0 mg/kg/day administered orally or via G-tube for up to 144 weeks.
  Interventions: Drug: PRAX-562

INTERVENTIONS:
Drug: PRAX-562 — Once daily oral or G-tube treatment.

SUMMARY:
A Clinical Trial of PRAX-562 in Subjects With Developmental and Epileptic Encephalopathies (DEE)

DETAILED DESCRIPTION:
A Phase 2, double-blind, randomized clinical trial to evaluate the safety and tolerability of PRAX 562 in pediatric participants with SCN2A- and SCN8A- DEEs.

ELIGIBILITY:
Inclusion Criteria:

* Has a documented variant in SCN2A with onset of seizures occurring in the first 3 months of life or has a diagnosis of SCN8A-DEE supported by both clinical and genetic findings.
* Has a seizure frequency as follows:

  * At least 8 countable motor seizures in the 4 weeks immediately prior to Screening as reported by the parent/legal guardian or in the opinion of the investigator as documented in medical notes.

AND o At least 8 countable motor seizures during the 28 day Baseline Observation Period (during which seizure frequency is recorded in a daily seizure diary).

• Additional inclusion criteria apply and will be assessed by the study team.

Exclusion Criteria:

* Has any clinically significant or known pathogenic or likely pathogenic genetic variant other than in SCN2A and SCN8A or a genetic variant that may explain or contribute to the participant's epilepsy and/or developmental disorder.
* Has a documented, functionally characterized loss-of-function (LoF) missense variant or a presumed LoF variant (nonsense or frameshift variant) based on genetic testing and/or clinical evidence that prior exposure to a sodium channel blocker (SCB) medication worsened seizures.
* Has 2 or more episodes of convulsive status epilepticus requiring hospitalization and intubation in the 6 months prior to Screening.
* Additional exclusion criteria apply and will be assessed by the study team.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
PART A (Cohorts 1 and 2) RDB: To evaluate the safety and tolerability of PRAX 562 in pediatric participants with SCN2A- and SCN8A- DEEs | 16 weeks
  Changes from baseline in monthly (28-day) motor seizure frequency
PART B (Cohorts 1 and 2) OLE: To evaluate the long-term safety and tolerability of PRAX-562 in pediatric participants with DEEs | 48 weeks
  Incidence and severity of TEAEs

SECONDARY OUTCOMES:
PART A (Cohorts 1 and 2) RDB: To assess the effect of PRAX-562 on the frequency of countable motor seizures in pediatric participants with DEEs | 16 weeks
  Changes from baseline in monthly (28-day) motor seizure frequency
Plasma concentrations of PRAX-562 | 16 weeks
  Sparse pharmacokinetic (PK) sampling will be used to calculate mean concentrations at baseline, and at Weeks 2, 4, 6, 8,10, 12 and 16.
Seizure Frequency (OLE Extension) | 48 weeks
  Efficacy assessments (seizure diary) will be collected daily and reviewed at timepoints Day 1, Week 16, Week 32, and Week 48.
To assess the effect of PRAX-562 on the frequency of countable motor seizures in pediatric participants with DEEs | 16 weeks
  Changes from baseline in monthly (28-day) motor seizure frequency
Incidence of Treatment-Emergent Adverse Events (TEAEs) [Safety and Tolerability]) | 16 weeks
  The number of participants with treatment-emergent adverse events will be reported by severity and preferred term.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Praxis Precision Medicines
Locations (8):
- United States (4):
  - Praxis Research Site, Atlanta, Georgia
  - Praxis Research Site, Chicago, Illinois
  - Praxis Research Site, Minneapolis, Minnesota
  - Praxis Research Site, Hackensack, New Jersey
- Praxis Research Site, Tel Litwinsky, Israel
- Praxis Research Site, Madrid, Spain
- United Kingdom (2):
  - Praxis Research Site, Glasgow
  - Praxis Research Site, London